CLINICAL TRIAL: NCT03217019
Title: Comparison of Radial Artery Cannulation Technique in Pediatric Patients: Direct Versus Guidewire-assisted
Brief Title: Guidewire-assisted Radial A-line in Neonate and Infant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Tae Kim, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1706-086-859
Record Dates: First submitted 2017-07-10; First posted 2017-07-13 (Actual); Last update posted 2019-04-08 (Actual); Status verified 2019-04

CONDITIONS: Arterial Line
Keywords: Radial Artery; Vascular Catheters

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Guidewire (Experimental): 1. Radial artery puncture with direct radial pulse palpation.
  2. 24G angiocatheter insertion with guidewire-assist. (Catheter over guidewire)
  Interventions: Procedure: Guidewire-assist
- Direct (Active Comparator): 1. Radial artery puncture with direct radial pulse palpation.
  2. 24G angiocatheter insertion without guidewire-assist. (Catheter over needle)
  Interventions: Procedure: Direct

INTERVENTIONS:
Procedure: Guidewire-assist — catheter insertion with guidewire-assist(catheter over guidewire)
  Arms: Guidewire
Procedure: Direct — catheter insertion without guidewire assist(catheter over needle)
  Arms: Direct

SUMMARY:
In neonate and infant, radial artery cannulation may be challenging and multiple attempts are required because of the small diameter.

The invastigators will compare the success rates of radial arterial cannulation with a guidewire-assisted technique and the direct technique in pediatric patient(<1yr).

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients undergoing general anesthesia with arterial cannulation (for hemodynamic monitoring or blood sampling)

Exclusion Criteria:

* Skin lesion, infection, hematoma, recent cannulation at cannulation site
* Unstable radial pulse (d/t unstable vital sign, or arrhythmias)

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2017-08-07 (Actual); Primary Completion 2018-07-04 (Actual); Study Completion 2018-07-04 (Actual)

PRIMARY OUTCOMES:
success rate at 1st attempt (%) | from arterial cannulation to successful invasive BP monitoring (up to 1 hour)
  successful catheter insertion after obtaining 1st blood flush in angiocatheter.

SECONDARY OUTCOMES:
total elapsed time (seconds) | from arterial cannulation to successful invasive BP monitoring (up to 1 hour)
  total time for successful cannulation.
number of total cannulation attempts (number) | from arterial cannulation to successful invasive BP monitoring (up to 1 hour)
  number of total attempts until successful cannulation. (1 attempt = 1 blood flush)
number of total catheter used (number) | from arterial cannulation to successful invasive BP monitoring (up to 1 hour)
  number of total catheter used until successful cannulation.
malfunction of arterial line | from the start of invasive BP monitoring until the end of anesthesia (up to 1 day)
  pressure monitoring, blood sampling
complications | from the arterial cannulation until the end of anesthesia (up to 1 day)
  hematoma, ischemia

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Tae Kim, MD, PhD, Study Chair — Professor
Locations (1):
- Jin-Tae Kim, Seoul, South Korea

REFERENCES:
- [Derived] Jang YE, Kim EH, Lee JH, Kim HS, Kim JT. Guidewire-assisted vs. direct radial arterial cannulation in neonates and infants: A randomised controlled trial. Eur J Anaesthesiol. 2019 Oct;36(10):738-744. doi: 10.1097/EJA.0000000000001064. PMID 31356376